CLINICAL TRIAL: NCT03382977
Title: A Three-part, Phase I/II Dose-Escalation Study to Define the Safety, Tolerability, and Optimal Dose of Candidate GBM Vaccine VBI-1901 With Subsequent Extension of Optimal Dose in Recurrent GBM Subjects
Brief Title: Study to Evaluate Safety, Tolerability, and Optimal Dose of Candidate GBM Vaccine VBI-1901 in Recurrent GBM Subjects
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VBI Vaccines Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VBI-1901-01
Record Dates: First submitted 2017-11-23; First posted 2017-12-26 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-07

CONDITIONS: Glioblastoma Multiforme
Keywords: GBM; Glioblastoma; eVLP; VBI-1901; vaccine; immunotherapy; CMV; CNS; Brain; Cancer
MeSH Terms: conditions — Glioblastoma; Neoplasms | interventions — Carmustine; Lomustine

STUDY DESIGN:
Intervention Model Description: 3+ 3 Dose Escalation
  Therapeutic Vaccine: VBI-1901
  The vaccine is formulated with GM-CSF adjuvant and administered intradermally (ID) or with AS01B adjuvant and administered intramuscularly (IM) to patients with recurrent GBM.
Masking Description: None, open-label Allocation (FDAAA)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Part A Dose Level 1 (Experimental): VBI-1901 low dose (0.4 μg pp65 content) vaccine formulated with GM-CSF (200 μg) in 0.2 mL volume, given in two equal intradermal injections
  Interventions: Biological: VBI-1901
- Part A Dose Level 2 (Experimental): VBI-1901 intermediate dose (2 μg pp65 content) vaccine formulated with GM-CSF (200 μg) in 0.2 mL volume, given in two equal intradermal injections
  Interventions: Biological: VBI-1901
- Part A Dose Level 3 (Experimental): VBI-1901 high dose (10 μg pp65 content) vaccine formulated with GM-CSF (200 μg) in 0.2 mL volume, given in two equal intradermal injections
  Interventions: Biological: VBI-1901
- Part B GM-CSF Adjuvant (Experimental): VBI-1901 10 μg HCMV pp65 formulated with GM-CSF (200 μg) in 0.2 to 0.4 mL volume, given in two to four equal ID injections.
  Interventions: Biological: VBI-1901
- Part B AS01B Adjuvant (Experimental): VBI-1901 10 μg HCMV pp65 formulated with AS01B (50 μg of QS-21 and 50 μg of MPL per dose) in 1.0 mL volume, given in one IM injection
  Interventions: Biological: VBI-1901
- Part C VBI-1901 with GM-CSF Adjuvant (Experimental): VBI-1901 10 μg HCMV pp65 formulated with GM-CSF (200 μg) in 0.2 mL volume, given in two equal ID injections.
  Interventions: Biological: VBI-1901
- Part C Standard of Care Treatment (Active Comparator): Single-agent standard-of-care (SOC) treatment with either carmustine intravenously at a dose of 150 mg/m² or lomustine orally at a dose of 110 mg/m² (up to a maximum dose of 200 mg).
  Interventions: Drug: Carmustine; Drug: Lomustine

INTERVENTIONS:
Biological: VBI-1901 — The vaccine is formulated with GM-CSF adjuvant and administered intradermally (ID) or with AS01B adjuvant and administered intramuscularly (IM) to patients with recurrent GBM.
  Arms: Part A Dose Level 1; Part A Dose Level 2; Part A Dose Level 3; Part B AS01B Adjuvant; Part B GM-CSF Adjuvant; Part C VBI-1901 with GM-CSF Adjuvant
Drug: Carmustine — Treatment with carmustine intravenously at a dose of 150 mg/m² on Day 1 and every 6 weeks until the earlier of disease progression or intolerable toxicity.
  Other Names: BiCNU
  Arms: Part C Standard of Care Treatment
Drug: Lomustine — Treatment with lomustine given orally at a dose of 110 mg/m² (up to a maximum dose of 200 mg) on Day 1 and every 6 weeks until the earlier of disease progression or intolerable toxicity.
  Other Names: Gleostine
  Arms: Part C Standard of Care Treatment

SUMMARY:
The purpose of this study is to assess the safety and tolerability of VBI-1901 in subjects with recurrent malignant gliomas (glioblastoma, or GBM).

DETAILED DESCRIPTION:
This is a three-part, dose-escalation study to define the safety, tolerability, and optimal dose level of candidate GBM vaccine VBI-1901 with subsequent extension of optimal dose level in recurrent GBM subjects and comparison with standard of care (SOC) treatment. Subjects in groups receiving VBI-1901 vaccination will continue to receive vaccine every 4 weeks until tumor progression per immunotherapy Response Assessment for Neuro-Oncology (iRANO)/Response Assessment for Neuro-Oncology (RANO) criteria.

ELIGIBILITY:
PART A DOSE ESCALATION

Inclusion Criteria: Part A Dose Escalation

1. 18-70 years of age
2. Histologically confirmed WHO grade IV glioblastoma
3. Unequivocal evidence of a tumor recurrence (any number of recurrences) or progression after an initial treatment regimen (prior to enrollment on this study) as assessed by MRI of the brain with and without contrast within 30 days prior to the initiation of injections of VBI-1901. An initial therapy requires surgery and radiation therapy, with or without temozolomide. In addition, alternate therapy (with or instead of temozolomide) is permitted as part of initial therapy.
4. Recovery from the effects of surgery.
5. Corticosteroid (dexamethasone or equivalent) dosage ≤ 4mg daily that has been stable or decreasing for at least 5 days.
6. Recovery from prior therapy toxicity defined as resolution of all treatment-related adverse events (AEs) to Grade ≤ 1 or pre-treatment baseline (except alopecia).
7. Karnofsky performance status (KPS) score ≥ 70%.
8. Adequate organ function, including the following:

   1. Absolute neutrophil count (ANC) ≥ 1,000/μL, platelets ≥ 100,000/μL
   2. Serum creatinine < 1.5 × the upper limit of normal (ULN)
   3. Bilirubin < 1.5 × ULN
   4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 × ULN
9. Women of childbearing potential: negative urine pregnancy test within 14 days prior to the start of VBI-1901 treatment.
10. Female subjects of childbearing potential and sexually active male subjects must agree to use an acceptable form of contraception for heterosexual activity (i.e., oral contraceptives, double barrier methods, hormonal injectable, transdermal, or implanted contraceptives, tubal ligation, or vasectomy of their sexual partner(s) for >30 days before Screening, during the study, and for 60 days after the last dose of study drug).
11. Female subjects without childbearing potential (spontaneous amenorrhea for > 12 months or surgically sterilized by tubal ligation, hysterectomy, or bilateral oophorectomy > 6 months before Screening) are eligible for inclusion without contraceptive use restriction.
12. Able and willing to comply with protocol requirements in the opinion of the Investigator, including being able to have an MRI.
13. Written consent has been obtained.
14. Tumor specimen available for central pathological review.

Exclusion Criteria: Part A Dose Escalation

1. Contrast-enhancing residual tumor that is associated with either diffuse sub-ependymal or leptomeningeal dissemination.
2. Requirement of systemic corticosteroid therapy > 4 mg/day of dexamethasone or equivalent or requirement of increasing dose of systemic corticosteroids during the 7 days prior to the start of VBI-1901 treatment.
3. Evidence of HCMV viremia in serum of > 18,200 (4.3Log10) IU/mL using FDA approved COBAS® AmpliPrep/COBAS® TaqMan® HCMV test (Roche).
4. Surgical resection or major surgical procedure within 4 days prior to the start of VBI-1901, or stereotactic biopsy within 7 days prior to the start of VBI-1901.
5. Active infection requiring intravenous antibiotics or antiviral.
6. History of cancer (other than GBM or prostate) within the past 2 years that could negatively impact survival and/or potentially confound tumor response assessments within this study.
7. Known immunosuppressive disease or active systemic autoimmune disease such as systemic lupus erythematosus, human immunodeficiency virus infection, Hepatitis B virus or Hepatitis C virus infections. Subjects with vitiligo, type 1 diabetes mellitus, hypothyroidism due to autoimmune condition only requiring hormone replacement therapy, psoriasis not requiring systemic therapy, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
8. Immunosuppressive agent within 4 weeks prior to the start of VBI-1901 treatment.
9. Evidence of intra-tumoral or peri-tumoral hemorrhage on baseline, other than those that are ≤Grade 1 and either post-operative or stable on at least 2 consecutive MRI scans.
10. Any condition which in the investigator's opinion makes the subject unsuitable for study participation.
11. Lack of family or social support structure that would preclude continued participation in the study.

PART B OPTIMAL DOSE

Inclusion Criteria: Part B Optimal Dose

1. 18-70 years of age.
2. Histologically confirmed WHO grade IV glioblastoma.
3. Unequivocal evidence of a first tumor recurrence with measurable disease, of an area no greater than 400 mm2, which may include patients with resected first recurrence tumor after an initial treatment regimen (prior to enrollment on this study) consisting of surgical intervention (tumor resection) and radiation, with or without temozolomide chemotherapy (depending on the MGMT methylation status), as assessed by MRI of the brain with and without contrast within 30 days prior to the initiation of injections of VBI-1901. In addition, alternate chemotherapy (with or instead of temozolomide) is permitted as part of initial therapy.
4. At least 12 weeks since radiotherapy treatment and/or 23 days after chemotherapy prior to first dose of VBI-1901.
5. Recovery from the effects of surgery.
6. Corticosteroid (dexamethasone or equivalent) dosage ≤ 4mg daily that has been stable or decreasing for at least 5 days.
7. Recovery from prior therapy toxicity, defined as resolution of all treatment-related adverse events (AEs) to Grade ≤ 1 or pre-treatment baseline (except alopecia).
8. Karnofsky performance status (KPS) score ≥ 70%.
9. Adequate organ function, including the following:

   1. Absolute neutrophil count (ANC) ≥ 1,000/μL, platelets ≥ 100,000/μL; absolute lymphocyte count ≥ 500/uL;
   2. Serum creatinine < 1.5 × the upper limit of normal (ULN);
   3. Bilirubin < 1.5 × ULN;
   4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 × ULN.
10. Women of childbearing potential must have a negative urine pregnancy test within 14 days prior to the start of VBI-1901 treatment.
11. Female subjects of childbearing potential and sexually active male subjects must agree to use an acceptable form of contraception for heterosexual activity (i.e., oral contraceptives, double barrier methods, hormonal injectable, transdermal, or implanted contraceptives, tubal ligation, or vasectomy of their sexual partner(s) for > 30 days before Screening, during the study, and for 60 days after the last dose of study drug).
12. Female subjects without childbearing potential (spontaneous amenorrhea for > 12 months or surgically sterilized by tubal ligation, hysterectomy, or bilateral oophorectomy > 6 months before Screening) are eligible for inclusion without contraceptive use restriction.
13. Able and willing to comply with protocol requirements, in the opinion of the Investigator.
14. Written consent has been obtained.
15. Tumor specimen available for central pathological review.

Exclusion Criteria: Part B Optimal Dose

1. Contrast-enhancing residual tumor that is any of the following:

   1. An area greater than 400mm2;
   2. Multi-focal (defined as two separate areas of contrast enhancement measuring at least 1 cm in 2 planes that are not contiguous on either fluid-attenuated inversion recovery (FLAIR) or T2 sequences);
   3. Associated with either diffuse sub-ependymal or leptomeningeal dissemination.
2. IDH1/2 has been proven to be mutated by IHC or PCR or if recurrent GBM was previously a lower grade glioma and wildtype IDH1/2 status has not been confirmed.
3. Requirement of systemic corticosteroid therapy > 4 mg/day of dexamethasone or equivalent or requirement of increasing dose of systemic corticosteroids during the 7 days prior to the start of VBI-1901 treatment.
4. Evidence of HCMV viremia in plasma of >18,200 (4.3log10) IU/mL using FDA approved COBAS® AmpliPrep/COBAS® TaqMan® HCMV test (Roche).
5. Prior treatment involving immunotherapy, including oncolytic viruses, therapeutic vaccination, or biologics (e.g. monoclonal antibodies, such as bevacizumab) presumed to have immunomodulatory effects.
6. Surgical resection or major surgical procedure within 14 days prior to the start of VBI-1901, or stereotactic biopsy within 14 days prior to the start of VBI-1901.
7. Radiation therapy, local therapy (except for surgical re-resection), or systemic therapy following first recurrence/progressive disease. Excluded local therapies include stereotactic radiation boost, implantation of carmustine biodegradable wafers (Gliadel), intratumoral or convection- enhanced delivery administered agents, etc.
8. Concurrent therapy with Optune® or use within 1 week of start of treatment with VBI-1901.
9. Active infection requiring intravenous antibiotics or antivirals.
10. History of cancer (other than GBM or prostate) within the past 2 years that has metastatic or local recurrence potential and could negatively impact survival and/or potentially confound tumor response assessments within this study.
11. Known immunosuppressive disease or active systemic autoimmune disease such as systemic lupus erythematosus, human immunodeficiency virus infection, Hepatitis B virus or Hepatitis C virus infections. Subjects with vitiligo, type 1 diabetes mellitus, hypothyroidism due to autoimmune condition only requiring hormone replacement therapy, psoriasis not requiring systemic therapy, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
12. Immunosuppressive agent within 4 weeks prior to the start of VBI-1901 treatment.
13. Any severe adverse event or allergy suspected or attributed to the shingles vaccines that contains AS01B components.
14. Evidence of intra- or peri-tumoral hemorrhage on baseline MRI scan, other than those that are ≤Grade 1 and either post-operative or stable on at least 2 consecutive MRI scans.
15. Any condition which in the investigator's opinion makes the subject unsuitable for study participation.
16. Lack of family or social support structure that would preclude continued participation in the study.

PART C RANDOMIZED OPEN-LABEL STUDY EXTENSION

INCLUSION CRITERIA

1. 18 years of age or older (no age upper limit).
2. Histologically confirmed supratentorial 2016 WHO classification grade IV Glioblastoma, IDH-wildtype or grade 4 in the 2021 WHO classification. Tumors that are histologically lower grade but are classified as glioblastoma using the WHO 2021 criteria because of molecular alterations (TERT promoter mutation and/or EGFR amplification and/or combined chromosome 7 gain/10 loss) are not eligible.
3. Unequivocal evidence of a first tumor recurrence with measurable disease of an area no greater than 600 mm2, which may include patients with resected first recurrence tumor, after an initial treatment regimen (prior to enrollment on this study) consisting of surgical intervention (tumor resection) and radiation, with or without temozolomide chemotherapy (depending on the MGMT methylation status), as assessed by MRI of the brain with and without contrast completed within 30 days prior to screening visit, if not it should be performed as part of screening visit. In addition, alternate bio/chemotherapy (with or instead of temozolomide) other than nitrosourea is permitted as part of initial therapy.
4. At least 12 weeks since radiotherapy treatment and/or 23 days after chemotherapy prior to first dose of VBI-1901 or SOC treatment. Patients with recurrent GBM within 12 weeks of radiation therapy may be included if they have surgically proven tumor recurrence (i.e.

   this is proven to not be pseudoprogression).
5. Recovery from the effects of surgery.
6. Corticosteroid (dexamethasone or equivalent) dosage ≤ 2 mg daily that has been stable for at least 5 days before randomization into the study.
7. Recovery from prior therapy toxicity, defined as resolution of all treatment related adverse events (AEs) to Grade ≤ 1 or pre-treatment baseline (except alopecia).
8. Karnofsky performance status (KPS) score ≥70%.
9. Adequate organ function, including the following:

   1. Absolute neutrophil count (ANC) ≥ 1,000/μL, platelets ≥ 100,000/μL; Absolute lymphocyte count ≥ 500/uL; CD4/CD8 ratio ≥1 or CD4 count ≥ 400/uL;
   2. Serum creatinine < 1.5 × the upper limit of normal (ULN);
   3. Bilirubin < 1.5 × ULN;
   4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 × ULN.
10. Women of childbearing potential must have a negative urine pregnancy test within 21 days prior to the start of treatment.
11. Female subjects of childbearing potential and sexually active male subjects must agree to use an acceptable form of contraception for heterosexual activity (i.e., oral contraceptives, double barrier methods, hormonal injectable, transdermal, or implanted contraceptives, tubal ligation, or vasectomy of their sexual partner(s) for > 40 days before Screening, during the study, and for 60 days after the last dose of study drug).
12. Female subjects without childbearing potential (spontaneous amenorrhea for >12 months or surgically sterilized by tubal ligation, hysterectomy, or bilateral oophorectomy > 6 months before Screening) are eligible for inclusion without contraceptive use restriction.
13. Able and willing to comply with protocol requirements, in the opinion of the Investigator.
14. Written consent has been obtained.

EXCLUSION CRITERIA:

1. Contrast-enhancing residual tumor that is any of the following:

   1. An area greater than 600 mm2;
   2. Multicentric (defined as two separate areas of contrast enhancement measuring at least 1 cm in 2 planes that are not contiguous on either fluid-attenuated inversion recovery (FLAIR) or T2 sequences);
   3. Associated with either diffuse sub-ependymal or leptomeningeal dissemination.
2. If recurrent GBM was previously a lower grade glioma and wildtype IDH1/2 status has not been confirmed.
3. Requirement of systemic corticosteroid therapy > 2 mg/day of dexamethasone or equivalent during the 5 days prior to the start of treatment.
4. Evidence of HCMV viremia in plasma of > 18,200 (4.3log10) IU/mL using FDA approved COBAS® AmpliPrep/COBAS® TaqMan® HCMV test (Roche) or other qualified HCMV assay.
5. Prior treatment involving immunotherapy, including oncolytic viruses, therapeutic vaccination, or biologics presumed to have immunomodulatory effects. Prior bevacizumab therapy is allowed, requiring at least 28 days washout period before randomization.
6. Surgical resection or major surgical procedure within 14 days prior to the start of treatment, or stereotactic biopsy within 7 days prior to the start of treatment.
7. Radiation therapy, local therapy (except for surgical re-resection), or systemic therapy following first recurrence/progressive disease. Excluded local therapies include stereotactic radiation boost, implantation of carmustine biodegradable wafers (Gliadel), intratumoral or convectionenhanced delivery administered agents, etc.
8. More than 1 (one) line of prior chemotherapy (as an example, temozolomide given with radiotherapy and after radiotherapy before recurrence is considered a single line).
9. Concurrent therapy with Optune® or use within 1 week of start of treatment. Previous use of Optune® in the primary setting does not preclude participation in this clinical trial.
10. Active infection requiring intravenous antibiotics or antivirals.
11. History of cancer (other than GBM or prostate) within the past 2 years that has metastatic or local recurrence potential and could negatively impact survival and/or potentially confound tumor response assessments within this study.
12. Known immunosuppressive disease or active systemic autoimmune disease such as systemic lupus erythematosus, human immunodeficiency virus infection, Hepatitis B virus or Hepatitis C virus infections. Subjects with vitiligo, type 1 diabetes mellitus, hypothyroidism due to autoimmune condition only requiring hormone replacement therapy, psoriasis not requiring systemic therapy, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
13. Any known allergies to the ingredients of VBI-1901 or GM-CSF or carmustine or lomustine.
14. Evidence of intra- or peri-tumoral hemorrhage on baseline MRI scan, other than those that are ≤Grade 1 and either post-operative or stable on at least 2 consecutive MRI scans.
15. Any medical or social condition which in the investigator's opinion makes the subject unsuitable for study participation. For instance, lack of family or social support structure that would preclude continued participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2017-12-06 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) occurring during Part A of the study | Through 14 days after each study vaccination
Occurrence of AEs during each treatment cycle | Through 28 days after each study vaccination

SECONDARY OUTCOMES:
Serum antibody immune response | Baseline and 2 weeks after each dose of vaccine in Part A and Part B and every 3 months in Part C
  Assessment of IgG antibody to HCMV gB antigen by ELISA
Cellular immune responses | Baseline and 2 weeks after each dose of vaccine in Part A and Part B and every 3 months in Part C
  Assessment of IFN-γ and IL-5 positive peripheral blood mononuclear cells by ELISPOT
Progression free survival (PFS) | From the date of first dose to date of progression or death, as well as at 6, 12, 18 and 24 months
  Progression free survival (PFS) from date of first dose to date of progression (per iRANO/RANO criteria) or death, as well as at 6, 12, 18 and 24 months.
Overall survival (OS) | 6, 12, 18 and 24 months from date of first dose
Median overall survival in Part A and Part B of the study | Date of first dose to date of death from any cause, assessed up to 18 months
Reduction in steroid use compared to baseline | Baseline to study completion, an average of 12 months
Change in quality of life (QOL questionnaire) compared to baseline | Baseline to study completion, an average of 12 months
Tumor response rates (TRR) in Part C of the study | Baseline to study completion, an average of 12 months
  Complete response rate, partial response rate, progressive disease and stable disease
Safety and efficacy of VBI-1901 compared to standard of care (SOC) in Part C of study | Baseline to study completion, an average of 12 months
  An integrated analysis of safety and efficacy (OS, TRR, PFS) in subjects receiving VBI-1901 at 10 µg dose formulated with GM-CSF as compared to subjects receiving SOC

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Diaz-Mitoma, MD, Study Director — Variation Biotechnologies Inc.
Locations (12):
- United States (12):
  - University of California, Irvine, Irvine, California
  - University of California, San Diego, La Jolla, California
  - University of California, Los Angeles Neuro-Oncology Program, Los Angeles, California
  - Stanford, Stanford, California
  - Miami Cancer Institute, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - The Valley Hospital - Neurosurgeons of New Jersey, Ridgewood, New Jersey
  - The Neurological Institute of New York Columbia University Medical Center, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Providence - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes